CLINICAL TRIAL: NCT04757298
Title: Optimization of a New Adaptive Intervention to Increase COVID-19 Testing Among People at High Risk in an Urban Community
Brief Title: Optimization of a New Adaptive Intervention to Increase COVID-19 Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: North Jersey Community Research Initiative (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH); University of Michigan (Other)
Responsible Party: Principal Investigator, Liliane Cambraia Windsor, Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: UIUC-NJCRI 102497-18274-267805; 3R01MD010629-04S2 (NIH)
Record Dates: First submitted 2021-02-15; First posted 2021-02-17 (Actual); Results first posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: COVID-19 Testing
MeSH Terms: interventions — Referral and Consultation

STUDY DESIGN:
Intervention Model Description: SMART Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Navigation only (Other): Participants are randomized to receive navigation services only.
  Interventions: Behavioral: Navigation Services
- Navigation + Brief Counseling (Other): After initial randomization into NS, some participants are randomized to receive Brief Counseling (BC)
  Interventions: Behavioral: Navigation Services; Behavioral: Brief Counseling
- Navigation + Critical Dialogue (Other): After initial randomization into NS, some participants are randomized to receive Critical Dialogue (CD)
  Interventions: Behavioral: Navigation Services; Behavioral: Critical Dialogue
- Brochure only (Other): Participants are randomized to receive Brochure only.
  Interventions: Behavioral: Referral and Digital Brochure
- Brochure + Brief Counseling (Other): After initial randomization to receive a brochure, some participants are randomized to receive Brief Counseling (BC)
  Interventions: Behavioral: Brief Counseling; Behavioral: Referral and Digital Brochure
- Brochure + Critical Dialogue (Other): After initial randomization to receive a brochure, some participants are randomized to receive Critical Dialogue (CD)
  Interventions: Behavioral: Critical Dialogue; Behavioral: Referral and Digital Brochure

INTERVENTIONS:
Behavioral: Navigation Services — Navigation services include assessment and support with service referrals. Each participant will meet with a peer navigator in person or on Zoom Conferencing for 30 minutes to go over results from their social and health needs assessment that is retrieved from the baseline assessment. The navigator shares information about COVID-19, answers questions about testing, and makes referrals to other needed services
  Arms: Navigation + Brief Counseling; Navigation + Critical Dialogue; Navigation only
Behavioral: Critical Dialogue — Critical Dialogue includes three one-hour-long, open-group-sessions facilitated in person or online by a trained licensed facilitator. Group critical dialogue is prompted by thematic images developed by the NCCB to foster a deeper understanding of how systematic stigma, feelings of rage as victims of discrimination, and/or apathy may impact participants' beliefs and behaviors related to COVID-19 and empower participants to make critical choices to protect their health and the health of their communities.
  Arms: Brochure + Critical Dialogue; Navigation + Critical Dialogue
Behavioral: Brief Counseling — Brief Counseling is a 15-minute post-COVID-19 test session delivered by a trained licensed clinician in person or via Zoom Conferencing. In the session, the clinician shares the test results and offers recommendations and information about COVID-19 treatment and prevention.
  Arms: Brochure + Brief Counseling; Navigation + Brief Counseling
Behavioral: Referral and Digital Brochure — Referral will consist of a five-minute phone call where an outreach worker offers participants information about COVID-19 testing and encourages them to get tested within one week. A digital brochure containing NJ recommendations is e-mailed or texted to participants.
  Arms: Brochure + Brief Counseling; Brochure + Critical Dialogue; Brochure only

SUMMARY:
This study tests an adaptation of the HIV Continuum of Prevention, Care, and Treatment Framework (CoPCT) for use in tracking COVID-19 testing and follow-up in a medically and socially vulnerable population. This study uses an integrated research collaborative framework that facilitates dialogue among researchers, community members, and service providers as a tool for optimizing the adaptive intervention and will take place at the North Jersey Community Research Initiative (NJCRI)

DETAILED DESCRIPTION:
This study will use the Multiphase Optimization Strategy (MOST) to optimize an adaptive intervention that successfully navigates COVID-19 medically or socially vulnerable people through a continuum of prevention, care and treatment (CoPCT) modeled on the HIV CoPCT. The COVID-19 CoPCT starts with testing and continues with successful adherence to prevention or treatment guidelines to help prevent and/or treat COVID-19. The study will assess the effectiveness of Navigation Services compared to referrals in increasing COVID-19 testing and Brief Counseling in increasing adherence to the State of NJ recommendations for COVID-19 prevention and treatment. The study will also examine the effect of Critical Dialogue on testing behavior among people who decline to be tested for COVID-19. The investigators will develop decision rules about what evidence-based-interventions work best for what types of people (e.g., those who test right away, versus decliners) and in what period of the COVID-19 continuum. Finally, the study will shed light on factors associated with testing and adherence to NJ recommendations. Investigators will follow Community Based Participatory Research principles in implementing a sequential, multiple assignment randomized trial (SMART) design. Adjusting for possible 15% loss to follow-up, a total sample of 670 people who are medically and socially vulnerable to infection and poor outcomes with COVID-19 will be enrolled as the intent-to treat-sample. The investigators are confident that they can recruit this sample in Essex County, NJ based on their previous experience and because the parent study research team has established relationships with other service agencies in the community from which, in addition to NJCRI, research participants will be drawn. The primary outcome is completion of the COVID-19 test within one week of the first intervention session The study will include 3 stages in which participants will be randomized to one of two possible interventions as follows:

1. Eligible and consenting participants will be randomized to receive the first-stage intervention: Navigation Services (NS) or standard services (referral to testing and NJ digital information brochure after testing). The primary outcome is completion of the COVID-19 test within one week of the intervention session.
2. Those who get tested will be randomized to receive the second-stage intervention: continue with NS or standard treatment or switch to Brief Counseling (BC). The outcome will be adherence to NJ recommendations. For those testing positive, adherence means engaging in a 14-day quarantine, receiving medical care as needed and contact tracing. For those testing negative, adherence means social distancing and wearing masks.
3. Those who do not get tested will be randomized into their second-stage intervention to continue with NS or digital brochure or switch to Critical Dialogue (CD). The outcome will be completing COVID-19 testing within 1 week of the second stage intervention session. Those who complete the testing will then be randomized to either continue with NS or digital brochure or switch to BC. Those who do not get tested will be randomized to continued NS or digital brochure or switch to CD. The outcome will be adherence to NJ recommendations, as defined above. All variables will be measured using standardized measures selected from the National Institutes of Health (NIH) PhenX Toolkit.

For the primary aim of comparing effects of Navigation Services versus referral on testing behavior and NJ recommendations adherence, using standard sample size formula for difference of two proportions, a total sample size of 582 subjects is needed to have 80% power at α=0.05 to detect a 10% difference in proportions, assuming 70% in the referral group will complete testing and adhere to specific NJ recommendations. The 582 sample size has 85% to detect a difference of 15% in adherence rates to NJ recommendations between two interventions.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* having high risk to contract COVID or develop related complications
* able to speak English
* able and willing to provide informed consent.

Exclusion Criteria:

* under 18 years of age
* not at high risk to contract COVID or develop related complications
* unable to speak English
* unable and unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 668 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liliane Windsor, PhD, Principal Investigator — University of Illinois Urbana Champaign
Locations (1):
- North Jersey Community Research Initiative, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data can be shared upon request for research purposes and under a data sharing agreement.
Supporting Information: ICF, Analytic Code
Time Frame: Upon request after the study is complete
Access Criteria: Must sign a data sharing agreement

REFERENCES:
- [Derived] Lee CA, Gamino D, Lore M, Donelson C, Windsor LC. Use of research electronic data capture (REDCap) in a sequential multiple assignment randomized trial (SMART): a practical example of automating double randomization. BMC Med Res Methodol. 2023 Jul 6;23(1):162. doi: 10.1186/s12874-023-01986-6. PMID 37415099
- [Derived] Lee CA, Gamino D, Lore M, Donelson C, Windsor LC. Use of research electronic data capture (REDCap) in a sequential multiple assignment randomized trial (SMART): A practical example of automating double randomization. Res Sq [Preprint]. 2023 Feb 24:rs.3.rs-2573133. doi: 10.21203/rs.3.rs-2573133/v1. PMID 36865151
- [Derived] Windsor L, Benoit E, M Pinto R, Sarol J. Optimization of a new adaptive intervention using the SMART Design to increase COVID-19 testing among people at high risk in an urban community. Trials. 2022 Apr 14;23(1):310. doi: 10.1186/s13063-022-06216-w. PMID 35421999

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited into the study at the North Jersey Community Research Initiative (NJCRI), one of New Jersey's largest and most comprehensive HIV/AIDS community-based organization.
Groups:
- Stage 1: Navigation: Participants in this arm were randomized to receive Navigation Services for Stage 1
- Stage 2 Navigation Followed by Navigation: Participants in this arm were first randomized to receive Navigation Services in Stage 1 and then were randomized again to receive Navigation Services in Stage 2
  Navigation Services: Navigation services include assessment and support with service referrals. Each participant will meet with a peer navigator in person or on Zoom Conferencing for 30 minutes to go over results from their social and health needs assessment that is retrieved from the baseline assessment. The navigator shares information about COVID-19, answers questions about testing, and makes referrals to other needed services
- Stage 2: Navigation Followed by Brief Counseling: Participants in this arm were randomized into Navigation Services in Stage 1 then randomized into Brief Counseling in Stage 2.
  Brief Counseling: Brief Counseling is a 15-minute post-COVID-19 test session delivered by a trained licensed clinician in person or via Zoom Conferencing. In the session, the clinician shares the test results and offers recommendations and information about COVID-19 treatment and prevention.
- Stage 2: Navigation Followed by Critical Dialogue: Participants in this arm were first randomized to receive Navigation Services in Stage 1 then randomized to receive Critical Dialogue in Stage 2.
  Critical Dialogue: Critical Dialogue includes three one-hour-long, open-group-sessions facilitated in person or online by a trained licensed facilitator. Group critical dialogue is prompted by thematic images developed by the NCCB to foster a deeper understanding of how systematic stigma, feelings of rage as victims of discrimination, and/or apathy may impact participants' beliefs and behaviors related to COVID-19 and empower participants to make critical choices to protect their health and the health of their communities.
- Stage 1: Brochure: Participants in this group were randomized to receive a digital brochure in Stage 1.
  Referral and Digital Brochure: Referral will consist of a five-minute phone call where an outreach worker offers participants information about COVID-19 testing and encourages them to get tested within one week. A digital brochure containing NJ recommendations is e-mailed or texted to participants.
- Stage 2: Brochure Followed by Brochure: Participants in this group were randomized to receive a brochure in Stage 1 and randomized to receive a brochure in Stage 2.
  Referral and Digital Brochure: Referral will consist of a five-minute phone call where an outreach worker offers participants information about COVID-19 testing and encourages them to get tested within one week. A digital brochure containing NJ recommendations is e-mailed or texted to participants.
- Stage 2: Brochure Followed by Brief Counseling: Participants in this group were randomized to receive a brochure in Stage 1 and randomized to receive Brief Counseling in Stage 2
  Brief Counseling: Brief Counseling is a 15-minute post-COVID-19 test session delivered by a trained licensed clinician in person or via Zoom Conferencing. In the session, the clinician shares the test results and offers recommendations and information about COVID-19 treatment and prevention.
- Stage 2: Brochure Followed by Critical Dialogue: Participants in this group were randomized to receive a Brochure in Stage 1 and randomized to receive Critical Dialogue in Stage 2.
  Critical Dialogue: Critical Dialogue includes three one-hour-long, open-group-sessions facilitated in person or online by a trained licensed facilitator. Group critical dialogue is prompted by thematic images developed by the NCCB to foster a deeper understanding of how systematic stigma, feelings of rage as victims of discrimination, and/or apathy may impact participants' beliefs and behaviors related to COVID-19 and empower participants to make critical choices to protect their health and the health of their communities.
Period: Stage 1: First Intervention
Arm/Group | Stage 1: Navigation | Stage 2 Navigation Followed by Navigation | Stage 2: Navigation Followed by Brief Counseling | Stage 2: Navigation Followed by Critical Dialogue | Stage 1: Brochure | Stage 2: Brochure Followed by Brochure | Stage 2: Brochure Followed by Brief Counseling | Stage 2: Brochure Followed by Critical Dialogue
Started (In Stage 1, participants were randomized to receive either Navigation Services or a Digital Brochure) | 328 | 0 | 0 | 0 | 340 | 0 | 0 | 0
Completed | 160 | 0 | 0 | 0 | 165 | 0 | 0 | 0
Not Completed | 168 | 0 | 0 | 0 | 175 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Stage 1: Navigation | Stage 2 Navigation Followed by Navigation | Stage 2: Navigation Followed by Brief Counseling | Stage 2: Navigation Followed by Critical Dialogue | Stage 1: Brochure | Stage 2: Brochure Followed by Brochure | Stage 2: Brochure Followed by Brief Counseling | Stage 2: Brochure Followed by Critical Dialogue
Started (After initial randomization into either Navigation or Brochure in Stage 1, participants were again randomized to receive Brief Counseling or Critical Dialogue in Stage 2) | 0 (This arm pertains to Stage 1 only) | 160 | 36 | 126 | 0 (This arm pertains to Stage 1 only.) | 165 | 32 | 137
Completed | 0 | 96 (Completion data for 12 participants in this arm is missing) | 16 | 16 | 0 | 164 (Completion data for 1 participant in this arm are missing) | 19 | 19
Not Completed | 0 | 64 | 20 | 110 | 0 | 1 | 13 | 118

BASELINE CHARACTERISTICS:
Population: This represents the Stage 2 baseline analysis population.
Groups:
- Navigation (1)+ Navigation (2): Participants in this group were randomized in Stage 1 to receive Navigation Services and randomized to receive Navigation Services in Stage 2.
  Navigation Services: Navigation services include assessment and support with service referrals. Each participant will meet with a peer navigator in person or on Zoom Conferencing for 30 minutes to go over results from their social and health needs assessment that is retrieved from the baseline assessment. The navigator shares information about COVID-19, answers questions about testing, and makes referrals to other needed services
- Navigation (1) + Brief Counseling (2): Participants in this Group were randomized to receive Navigation services in Stage 1 and randomized to receive Brief Counseling in Stage 2.
  Brief Counseling: Brief Counseling is a 15-minute post-COVID-19 test session delivered by a trained licensed clinician in person or via Zoom Conferencing. In the session, the clinician shares the test results and offers recommendations and information about COVID-19 treatment and prevention.
- Navigation (1) + Critical Dialogue (2): Participants in this group were randomized to receive Navigation Services in Stage 1 and randomized to receive Critical Dialogue in Stage 2.
  Critical Dialogue: Critical Dialogue includes three one-hour-long, open-group-sessions facilitated in person or online by a trained licensed facilitator. Group critical dialogue is prompted by thematic images developed by the NCCB to foster a deeper understanding of how systematic stigma, feelings of rage as victims of discrimination, and/or apathy may impact participants' beliefs and behaviors related to COVID-19 and empower participants to make critical choices to protect their health and the health of their communities
- Brochure (1) + Brochure (2): Participants in this group were randomized in stage 1 to receive a digital brochure and randomized to receive a digital brochure in Stage 2.
  Referral and Digital Brochure: Referral will consist of a five-minute phone call where an outreach worker offers participants information about COVID-19 testing and encourages them to get tested within one week. A digital brochure containing NJ recommendations is e-mailed or texted to participants.
- Brochure (1)+ Brief Counseling (2): Participants in this group were randomized in Stage 1 to receive a Brochure and were randomized to receive Brief Counseling in Stage 2.
  Brief Counseling: Brief Counseling is a 15-minute post-COVID-19 test session delivered by a trained licensed clinician in person or via Zoom Conferencing. In the session, the clinician shares the test results and offers recommendations and information about COVID-19 treatment and prevention.
- Brochure (1) + Critical Dialogue (2): Participants in this group were randomized to receive Navigation Services in Stage 1 and were randomized to receive Critical Dialogue in Stage 2.
  Critical Dialogue: Critical Dialogue includes three one-hour-long, open-group-sessions facilitated in person or online by a trained licensed facilitator. Group critical dialogue is prompted by thematic images developed by the NCCB to foster a deeper understanding of how systematic stigma, feelings of rage as victims of discrimination, and/or apathy may impact participants' beliefs and behaviors related to COVID-19 and empower participants to make critical choices to protect their health and the health of their communities.
- Total: Total of all reporting groups
Arm/Group | Navigation (1)+ Navigation (2) | Navigation (1) + Brief Counseling (2) | Navigation (1) + Critical Dialogue (2) | Brochure (1) + Brochure (2) | Brochure (1)+ Brief Counseling (2) | Brochure (1) + Critical Dialogue (2) | Total
Number analyzed (Participants) | 160 | 36 | 126 | 165 | 32 | 137 | 656
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 153 | 34 | 122 | 159 | 30 | 132 | 630
  >=65 years | 7 | 2 | 4 | 6 | 2 | 5 | 26
Sex/Gender, Customized [Count of Participants; unit: Participants] — Self-report biological sex assigned at birth
  Participants
    Male | 86 | 25 | 68 | 90 | 19 | 76 | 364
    Female | 72 | 10 | 53 | 67 | 12 | 57 | 271
    none of these describe me (includes those identifying as non-binary, transgender, and bi-gender) | 2 | 1 | 5 | 7 | 0 | 4 | 19
    Gender Missing/Unknown | 0 | 0 | 0 | 1 | 1 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 4 | 17 | 25 | 4 | 24 | 96
  Not Hispanic or Latino | 133 | 30 | 105 | 133 | 23 | 105 | 529
  Unknown or Not Reported | 5 | 2 | 4 | 7 | 5 | 8 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants were asked to select all races that applied to them. Thus, summation of responses will not equate to the total analyzed sample.
  Participants
    American Indian or Alaskan Native | 10 | 0 | 7 | 7 | 1 | 8 | 33
    Native Hawaiian or Pacific Islander | 1 | 0 | 2 | 2 | 0 | 4 | 9
    Black or African American | 127 | 31 | 99 | 127 | 26 | 99 | 509
    Asian | 0 | 0 | 6 | 3 | 0 | 0 | 9
    White | 19 | 3 | 12 | 16 | 2 | 12 | 64
    Other or Unknown | 14 | 2 | 7 | 16 | 2 | 14 | 55
    Missing/Not Reported | 1 | 0 | 0 | 1 | 2 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 160 | 36 | 126 | 165 | 32 | 137 | 656
COVID tested within previous 30 days [Count of Participants; unit: Participants] — Participants reported they had taken a COVID test within the prior 30 days
  Participants | 40 | 12 | 26 | 40 | 8 | 39 | 165

OUTCOME MEASURES:

1. Primary Outcome: Stage 1: Completion of COVID-19 Test After First Randomization
Description: For the first stage intervention, the primary outcome is coming to the agency and completing the COVID-19 antigen test one week after completing the baseline.
Time Frame: Stage 1: Within one week of completing baseline.
Population: Population for Stage 1
Measure: Number; unit: participants
Groups:
- Navigation (1): Participants in this group are randomized to receive Navigation Services in Stage 1.
  Navigation Services: Navigation services include assessment and support with service referrals. Each participant will meet with a peer navigator in person or on Zoom Conferencing for 30 minutes to go over results from their social and health needs assessment that is retrieved from the baseline assessment. The navigator shares information about COVID-19, answers questions about testing, and makes referrals to other needed services
- Brochure Only: After initial randomization, some participants will be assigned to receive standard referral services. Those who complete the COVID-19 testing will again be randomized and some will receive a digital brochure.
  Referral and Digital Brochure: Referral will consist of a five-minute phone call where an outreach worker offers participants information about COVID-19 testing and encourages them to get tested within one week. A digital brochure containing NJ recommendations is e-mailed or texted to participants.
Arm/Group | Navigation (1) | Brochure Only
Number analyzed (Participants) | 328 | 340
participants
  Stage 1 COVID tested | 78 | 71
  Missing/Unknown | 0 | 0

2. Primary Outcome: Stage 2: Reported COVID Test in Last 30 Days at 6 Months Post Baseline
Description: For the second stage intervention, the primary outcome is self-reported completion of COVID-19 test in the past 30 days at the follow up completed 6 months after baseline. Study participants were asked whether they had completed a COVID-19 test in the past 30 days.
Time Frame: Stage 2: 6 months post baseline (4th follow up visit)
Population: Population includes baseline at Stage 2.
Measure: Number; unit: participants
Arm/Group | Navigation (1)+ Navigation (2) | Navigation (1) + Brief Counseling (2) | Navigation (1) + Critical Dialogue (2) | Brochure (1) + Brochure (2) | Brochure (1)+ Brief Counseling (2) | Brochure (1) + Critical Dialogue (2)
Number analyzed (Participants) | 160 | 36 | 126 | 165 | 32 | 137
participants
  Reported COVID tested in prior 30 days | 40 | 12 | 26 | 40 | 8 | 39
  Missing | 0 | 18 | 57 | 78 | 16 | 53

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline through follow up sessions (6 months)
Groups:
- Stage 1: Navigation: At Stage 1 randomization, participants were assigned to receive navigation services(NS).
  Navigation Services: Navigation services include assessment and support with service referrals. Each participant will meet with a peer navigator in person or on Zoom Conferencing for 30 minutes to go over results from their social and health needs assessment that is retrieved from the baseline assessment. The navigator shares information about COVID-19, answers questions about testing, and makes referrals to other needed services
- Stage 2: Navigation Followed by Navigation: After Stage 1 randomization to receive Navigation Services (NS) participants will again be randomized and continue receiving NS.
  Navigation Services: Navigation services include assessment and support with service referrals. Each participant will meet with a peer navigator in person or on Zoom Conferencing for 30 minutes to go over results from their social and health needs assessment that is retrieved from the baseline assessment. The navigator shares information about COVID-19, answers questions about testing, and makes referrals to other needed services
- Stage 2: Navigation Followed by Brief Counseling: After Stage 1 randomization to receive Navigation Services (NS), participants will again be randomized to receive Brief Counseling (BC)
  Brief Counseling: Brief Counseling is a 15-minute post-COVID-19 test session delivered by a trained licensed clinician in person or via Zoom Conferencing. In the session, the clinician shares the test results and offers recommendations and information about COVID-19 treatment and prevention.
- Stage 2: Navigation Followed by Critical Dialogue: After Stage1 randomization to receive Navigation Services (NS), participants will again be randomized and assigned to Critical Dialogue (CD)
  Critical Dialogue: Critical Dialogue includes three one-hour-long, open-group-sessions facilitated in person or online by a trained licensed facilitator. Group critical dialogue is prompted by thematic images developed by the NCCB to foster a deeper understanding of how systematic stigma, feelings of rage as victims of discrimination, and/or apathy may impact participants' beliefs and behaviors related to COVID-19 and empower participants to make critical choices to protect their health and the health of their communities.
- Stage 1: Brochure: At Stage 1 randomization, participants will be assigned to receive standard brochure services.
  Referral and Digital Brochure: Referral will consist of a five-minute phone call where an outreach worker offers participants information about COVID-19 testing and encourages them to get tested within one week. A digital brochure containing NJ recommendations is e-mailed or texted to participants.
- Stage 2: Brochure Followed by Brochure: After Stage 1 randomization to Brochure, participants will again be randomized and some will be assigned to again receive Brochure.
  Referral and Digital Brochure: Referral will consist of a five-minute phone call where an outreach worker offers participants information about COVID-19 testing and encourages them to get tested within one week. A digital brochure containing NJ recommendations is e-mailed or texted to participants.
- Stage 2: Brochure Followed by Brief Counseling: After Stage 1 randomization to Brochure, participants will again be randomized and some will be assigned to receive Brief Counseling (BC).
  Brief Counseling: Brief Counseling is a 15-minute post-COVID-19 test session delivered by a trained licensed clinician in person or via Zoom Conferencing. In the session, the clinician shares the test results and offers recommendations and information about COVID-19 treatment and prevention.
- Stage 2: Brochure Followed by Critical Dialogue: After Stage 1 randomization to Brochure, participants will again be randomized and some will be assigned to Critical Dialogue (CD).
  Critical Dialogue: Critical Dialogue includes three one-hour-long, open-group-sessions facilitated in person or online by a trained licensed facilitator. Group critical dialogue is prompted by thematic images developed by the NCCB to foster a deeper understanding of how systematic stigma, feelings of rage as victims of discrimination, and/or apathy may impact participants' beliefs and behaviors related to COVID-19 and empower participants to make critical choices to protect their health and the health of their communities.
Arm/Group | Stage 1: Navigation | Stage 2: Navigation Followed by Navigation | Stage 2: Navigation Followed by Brief Counseling | Stage 2: Navigation Followed by Critical Dialogue | Stage 1: Brochure | Stage 2: Brochure Followed by Brochure | Stage 2: Brochure Followed by Brief Counseling | Stage 2: Brochure Followed by Critical Dialogue
All-Cause Mortality (participants affected / at risk) | 0/328 | 0/160 | 0/36 | 0/126 | 0/340 | 0/165 | 0/32 | 0/137
Serious Adverse Events (participants affected / at risk) | 0/328 | 0/160 | 0/36 | 0/126 | 0/340 | 0/165 | 0/32 | 0/137
Other Adverse Events (participants affected / at risk) | 0/328 | 0/160 | 0/36 | 0/126 | 0/340 | 0/165 | 0/32 | 0/137

LIMITATIONS AND CAVEATS:
Note that 46% of the sample never completed follow-up 4.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-12-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT04757298/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT04757298/SAP_001.pdf
  • Informed Consent Form (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT04757298/ICF_002.pdf